CLINICAL TRIAL: NCT06913569
Title: Endobronchial Ultrasound-Guided Transtunnel Forceps Biopsy vs. Transbronchial Needle Aspiration for Diagnosing Inadequate Lymph Node Specimens Based on Macroscopic On-site Evaluation: A Prospective, Randomized, Multicenter Study
Brief Title: EBUS-TTFB vs EBUS-TBNA for Diagnosing Inadequate Lymph Node Specimens Based on MOSE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Jiayuan Sun, Director, Department of Respiratory Endoscopy, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: SHCHE202502
Record Dates: First submitted 2025-03-30; First posted 2025-04-06 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Lymphadenopathy
MeSH Terms: conditions — Lymphadenopathy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EBUS-TBNA (Active Comparator): Specimens were obtained using a 22-gauge biopsy needle by bronchoscope. Each lymph node was operated 4 passes.
  Interventions: Procedure: EBUS-TBNA
- EBUS-TTFB via a tunnel (Experimental): A tunnel to reach the lymph node is established by making use of a puncture dilation catheter, and specimens were obtained using a 1.5 mm biopsy forceps by bronchoscope. Conduct biopsies until 5-10 specimens are obtained, and the actual number of passes and effective specimens should be recorded.
  Interventions: Procedure: EBUS-TTFB

INTERVENTIONS:
Procedure: EBUS-TBNA — Participants with lymphadenopathy would receive EBUS-TBNA attempts to conduct diagnoses.
  Arms: EBUS-TBNA
Procedure: EBUS-TTFB — Participants with lymphadenopathy would receive EBUS-TTFB attempts to conduct diagnoses.
  Arms: EBUS-TTFB via a tunnel

SUMMARY:
The study aims to compare the efficacy and safety of endobronchial ultrasound-guided transtunnel forceps biopsy to transbronchial needle aspiration in diagnosing inadequate lymph node specimens based on macroscopic on-site evaluation.

DETAILED DESCRIPTION:
Mediastinal and hilar lymphadenopathy are common clinical conditions. Endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA) is the standard method recommended by guidelines for obtaining tissue from these patients. Endobronchial ultrasound-guided transbronchial forceps biopsy (EBUS-TBFB) can overcome the limitations of inadequate tissue acquisition with EBUS-TBNA, and its efficacy and safety have been proved. However, EBUS-TBFB often requires the assistance of the electrocautery for mediastinal window creation, which increases technical difficulty and requires electrosurgical equipment, making it unsuitable for application in grassroots hospitals.

This study aims to use the endobronchial ultrasound-guided transtunnel forceps biopsy (EBUS-TTFB) method. A single-use bronchoscopic puncture dilation catheter will be employed to establish a tunnel between the airway and the lymph node, with both puncture and dilation completed in the same procedure. Currently, there is a lack of prospective randomized controlled trials to verify the efficacy and safety of EBUS-TTFB.

This study is designed as a prospective, multicenter, randomized controlled trial. A total of 162 patients will be randomly allocated in a 1:1 ratio to the EBUS-TBNA group or the EBUS-TTFB group. The primary endpoint is thediagnostic yield. The secondary endpoints include specimen adequacy, procedure duration, tunnel creation success rate, and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Chest imaging shows mediastinal or hilar lymphadenopathy (short axis ≥10 mm), requiring EBUS-TBNA for definitive diagnosis;
3. EBUS-TBNA can be performed on these lymph nodes, and the specimens obtained from conventional EBUS-TBNA with three needle passes are inadequate (macroscopic visible core < 30 mm);
4. Willing to participate in this clinical study and sign the informed consent form.

Exclusion Criteria:

1. Enlarged lymph nodes are identified as cystic or abscesses;
2. Severe coagulopathy, insufficient anticoagulants/antiplatelets withdraw time or bleeding diathesis (platelets<50*109/L, INR>1.3) that do not meet bronchoscopy requirements;
3. Other contraindications to bronchoscopy or transbronchial biopsy, such as severe cardiopulmonary insufficiency, intolerance to anesthesia, or endoscopic procedures;
4. Patients who have participated in another clinical trial within the past three months;
5. Vulnerable groups, such as pregnant women
6. Any other condition that the investigator considers inappropriate for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield | Six months after the procedure
  The diagnostic yield is defined as the proportion of lymph nodes diagnosed by each biopsy to the total number of lymph nodes enrolled in the study.

SECONDARY OUTCOMES:
Sample adequacy | Six months after the procedure
  The adequacy rate of samples for genetic testing: measured as the percentage of lymph node samples qualified for next-generation sequencing among all malignant lymph nodes.
Total procedure time | During the procedure
  The total procedure time is defined as the time from the insertion of the bronchoscope to its removal.
TTFB procedure time | During the procedure
  The EBUS-TTFB procedure time is defined as the time from the insertion of the biopsy needle into the bronchoscope to the cessation of bleeding after the final TTFB.
TBNA procedure time | During the procedure
  The EBUS-TBNA procedure time is defined as the time from the insertion of the biopsy needle into the bronchoscope to the cessation of bleeding after the final TBNA.
Tunnel creation success rate | During the procedure
  Defined as the percentage of lymph nodes in the EBUS-TTFB group where successful tunneling was achieved among the total number of lymph nodes.
Incidence of complications | Six months after the procedure
  Including pneumothorax, infection, mediastinal hematoma, emphysema and etc.

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Sun, Study Director — Shanghai Chest Hospital
Locations (3):
- China (3):
  - The Fourth Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Shanghai Chest Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Huzhou Central Hospital, Huizhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No